CLINICAL TRIAL: NCT04709809
Title: Analysis of Retinal Vessel Pulsations With Electrocardiographic Gating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01036
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Vessels; Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: Data driven analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Measurement RVA / IOP / with ECG gating
  Interventions: Device: Retinal Vessel Analyzer recordings with electrocardiographic (ECG) gating

INTERVENTIONS:
Device: Retinal Vessel Analyzer recordings with electrocardiographic (ECG) gating — Video recordings of ocular fundus, an analysis of dynamic vessel diameters and putting them in ECG context.

SUMMARY:
Analysis of Retinal Vessel Analyzer (RVA) recordings of retinal vessel pulsations, and putting them in context of intraocular pressure (IOP) pulsations by means of electrocardiographic (ECG) gating, in order to determine the lead source for pulsations of retinal veins.

DETAILED DESCRIPTION:
Rationale / Objective is to construct the retinal vessels wall pulsation cycle using an electrocardiographic gating, and to analyse it in comparison with an analogue intraocular pressure (IOP) cycle.

Based on the amplitude and on the phase shift of pulsations of retinal vessel wall, the goal is to identify a lead source of the retinal venous pulsations (IOP pulsations, or alternative sources, e.g. cerebrospinal fluid pulsations).

Subjects will be recruited from the environment of the master thesis medical students, colleagues and friends and the informed consent will be handed to them personally. Exclusion criteria will be addressed. One random eye per subject will be selected. On the study day, first the mydriasis drops - phenylephrine + tropicamide - will be applied, then ECG electrodes attached; 20 minutes after the mydriasis drops, the first set of measurements will be performed: RVA recording with ECG gating, and Pascal Dynamic Contour Tonometry (DCT) recording with ECG gating. Ten minutes after this measurements, 100% oxygen 5 liters/min through nasal cannula will be applied for 2 minutes and then the same measurements repeated. Approximate time needed for the whole run - around 60 minutes per subject, including (dis)mounting the ECG electrodes and the mydriasis time.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Known ophthalmological disease, in particular vascular disease.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Phase shift between pulsations | day 1
  No phase shift versus phase shift between the venous amplitude maximum and the IOP pulsation maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Basel, Baseö, Switzerland

IPD SHARING:
Plan to Share IPD: No